CLINICAL TRIAL: NCT07314424
Title: The Effect of Preoperative Intravenous Ferric Derisomaltose and EPO and Tranexamic Acid Versus Usual Treatment in Patients With Preoperative Anemia or Iron Deficiency in Bone Tumor: a Single-center, Prospective, Open-label, RCT Study
Brief Title: The Effect of Preoperative Intravenous Ferric Derisomaltose and EPO and Tranexamic Acid in Patients With Preoperative Anemia or Iron Deficiency in Bone Tumor
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tang Xiaodong (Other)
Responsible Party: Sponsor-Investigator, Tang Xiaodong, professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-anemia-001
Record Dates: First submitted 2025-09-28; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Anemia
Keywords: anemia; bone tumor; perioperative; Blood management
MeSH Terms: conditions — Anemia; Bone Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isomaltose Anhydride Iron Group (Experimental): Calculate the patient's iron requirement based on a simplified scale for the isomaltose iron group; Yibiao 150IU/kg subcutaneous injection, no treatment in the conventional treatment group; 0.5g of tranexamic acid is administered locally after dilution before surgical closure
  Interventions: Drug: isomaltose iron
- Conventional treatment group (No Intervention): Traditional symptomatic treatment

INTERVENTIONS:
Drug: isomaltose iron — Calculate the patient's iron requirement based on a simplified scale for the isomaltose iron group; Yibiao 150IU/kg subcutaneous injection, no treatment in the conventional treatment group; 0.5g of tranexamic acid is administered locally after dilution before surgical closure
  Arms: Isomaltose Anhydride Iron Group

SUMMARY:
The pelvis and spine are common sites of primary and secondary bone tumors, and most patients require surgical treatment. However, due to bleeding, high tumor burden, and other reasons, iron deficiency anemia (IDA) is common in these patients. At present, allogeneic blood resources are scarce in China and even globally, and cancer patients cannot undergo autologous blood transfusion. In addition, there is a large amount of bleeding during pelvic and spinal open surgery, which collectively leads to a high incidence of perioperative anemia in patients with pelvic and spinal tumors, and even the loss of surgical opportunities. Therefore, perioperative blood management for bone tumor surgery is extremely important. The combination of intravenous iron and EPO has been proven to rapidly improve the hemoglobin levels of perioperative surgical patients in previous studies, but there is currently no research related to bone tumors. This study uses a single center, prospective, open label, randomized controlled clinical trial to explore the effects of preoperative application of intravenous isomaltose iron combined with erythropoietin and tranexamic acid compared to conventional treatment in patients with preoperative anemia or iron deficiency in bone tumor surgery, hoping to establish a standard paradigm for perioperative blood management in bone tumor patients.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 and above with primary malignant bone tumors and bone metastases who plan to undergo open surgery for the sacrum, pelvis, and spine.
* 5 ± 2 days before surgery, hemoglobin<130g/L, or iron deficiency (TSAT<20%)
* Patients are able to understand the research content and sign informed consent forms

Exclusion criteria:

Meet any of the following criteria;

* Ferritin>800 ng/ml or hemoglobin<70 g/L
* Expected survival period less than six months
* Women who are pregnant, breastfeeding, or planning to conceive
* Known to have allergic reactions to other iron agents
* Severe bone marrow suppression event (4th degree bone marrow suppression) occurred 4 weeks before enrollment
* Decompensated stage of liver disease
* Patients with combined acute phase infections
* Chronic kidney disease stage 3-5
* Patients who received oral iron, intravenous iron, EPO, or blood transfusion treatment within one month prior to the start of the study.
* Researchers believe that other conditions that are not suitable for participation in this study, such as deafness, Parkinson's disease, communication disorders, etc
* Participated in other clinical trials within the three months prior to participating in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Hb levels 21 days after surgery | Day 21

SECONDARY OUTCOMES:
Blood transfusion rate within 21 days after surgery | Day 21
Hb levels 14 days after surgery | Day 14

IPD SHARING:
Plan to Share IPD: Yes